CLINICAL TRIAL: NCT03185169
Title: GSM (Genitourinary Syndrome Of Menopause) Management In Breast Cancer Survivors
Acronym: GSM
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study design change required protocol/ICF changes, deemed more appropriate to terminate study and apply knowledge gained to potential future study design
Sponsor: Alta Bates Summit Medical Center (Other)
Responsible Party: Principal Investigator, Uma Suryadevara, MD, Alta Bates Summit Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GSM
Record Dates: First submitted 2017-05-26; First posted 2017-06-14 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Genitourinary Abnormality; Breast Cancer Female; Vaginal Abnormality; Urinary Tract Infections; Dyspareunia; Dysuria
Keywords: breast cancer survivor; postmenopausal; dysuria; dyspareunia; vaginal dryness; urinary tract infections; urinary frequency; urinary urgency; genital burning; genital itching; genital dryness
MeSH Terms: conditions — Urogenital Abnormalities; Urinary Tract Infections; Dyspareunia; Dysuria | interventions — Replens; Coconut Oil

STUDY DESIGN:
Intervention Model Description: Observational, prospective open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Replens and coconut oil (Other): Commercially available Replens applied via prefilled applicator into the vagina and coconut oil applied at the vaginal introitus and vulva. Both are to be administered by the patient 2 times per week, interval between dosing to be approximately 2 days. Patients will be encouraged to apply Preseed, coconut oil, or patient's personal lubricant of choice into the vagina prior to sexual activity.
  Interventions: Combination Product: Replens and coconut oil

INTERVENTIONS:
Combination Product: Replens and coconut oil

SUMMARY:
The impact of treatment for GSM on the quality of life will be examined for postmenopausal women (defined as last menstrual period > 1 year ago or 6 months ago with FSH >40) who have been diagnosed with breast cancer.

DETAILED DESCRIPTION:
Postmenopausal breast cancer survivors who report at least one GSM sign or symptom will be offered participation in an observational, prospective open label trial. Study duration will be 6 months.

Evidence of GSM symptoms will be evaluated by a board certified gynecologist. Upon satisfying the prescreen requirements, the patient's information will be forwarded to the sub-investigator, who will confirm study eligibility and make the final determination verifying the diagnosis of GSM. Participants will be using commercially available Replens applied via prefilled applicator into the vagina and coconut oil applied at the vaginal introitus and vulva. Both are to be administered by the patient 2 times per week, interval between dosing to be approximately 2 days. Patients will be encouraged to apply Preseed, coconut oil, or patient's personal lubricant of choice into the vagina prior to sexual activity. Patients will record dosing on the Intake Diary. Outcome measures will include:

Quality of Life DIVA (Day-to-Day Impact of Vaginal Aging) questionnaire will be administered at Baseline, at month 1, 3 and month 6. The FSFI (Female Sexual Function Index) questionnaire will also be used for sexually active patients at the same time points. This is an exploratory investigation. A planned paired T test will be applied to analyze the outcome and regroup after data has been collected on the first 14 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Postmenopausal women (defined as last menstrual period > 1 year ago or 6 months ago with FSH >40) who have been diagnosed with breast cancer including in situ carcinoma (DCIS, LCIS)
3. Have self-identified GSM signs and objective symptoms on baseline screening
4. Patients already using Replens™ or coconut oil will have a two week washout period prior to starting study treatment.
5. Medical History review and Pelvic Exam by a board certified gynecologist for baseline assessment OR medical records review by a board certified gynecologist or delegated study staff to confirm diagnosis of GSM. If GSM is to be verified by medical record review, the sub-investigator will make the final determination of eligibility.

Exclusion Criteria:

1. Use of any estrogen containing product within 4 weeks prior to screening
2. Endometrial hyperplasia, endometrial cancer, or other gynecologic malignancy
3. Patients with non GSM related signs and symptoms as verified by a board certified gynecologist will be excluded.
4. Any concurrent illness or disorder that, per the opinion of the investigator, would preclude the patient from meeting the study requirements.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Estimated)
Dates: Start 2016-11-18 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
Improvement of GSM signs and/or symptoms | 1 month
  To show improvement of GSM signs and/or symptoms at month 1 compared to baseline period of administration of the study intervention. This will be measured by administering the Quality of Life DIVA (Day-to-Day Impact of Vaginal Aging) questionnaire.
Improvement of GSM signs and/or symptoms | 3 months
  To show improvement of GSM signs and/or symptoms at month 3 compared to baseline period of administration of the study intervention. This will be measured by administering the Quality of Life DIVA (Day-to-Day Impact of Vaginal Aging) questionnaire.
Improvement of GSM signs and/or symptoms | 6 months
  To show improvement of GSM signs and/or symptoms at month 6 compared to baseline period of administration of the study intervention. This will be measured by administering the Quality of Life DIVA (Day-to-Day Impact of Vaginal Aging) questionnaire.

SECONDARY OUTCOMES:
Sexual health of breast cancer survivors who are sexually active who are enrolled in this study | 6 months
  This study will investigate the sexual health of breast cancer survivors who are sexually active and using Replens™, Preseed™, coconut oil, or the patient's personal lubricant of choice prior to intercourse by the FSFI (Female Sexual Function Index) questionnaire. The percent change, from baseline to 6 months, in painful sexual activity will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Uma Suryadevara, MD, Principal Investigator — Alta Bates Summit Medical Center
Locations (1):
- Alta Bates Summit Medical Center, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang AJ, Gregorich SE, Kuppermann M, Nakagawa S, Van Den Eeden SK, Brown JS, Richter HE, Walter LC, Thom D, Stewart AL. Day-to-Day Impact of Vaginal Aging questionnaire: a multidimensional measure of the impact of vaginal symptoms on functioning and well-being in postmenopausal women. Menopause. 2015 Feb;22(2):144-54. doi: 10.1097/GME.0000000000000281. PMID 24983271
- [Background] Davila GW, Singh A, Karapanagiotou I, Woodhouse S, Huber K, Zimberg S, Seiler J, Kopka SL. Are women with urogenital atrophy symptomatic? Am J Obstet Gynecol. 2003 Feb;188(2):382-8. doi: 10.1067/mob.2003.23. PMID 12592244
- [Background] Larmo PS, Yang B, Hyssala J, Kallio HP, Erkkola R. Effects of sea buckthorn oil intake on vaginal atrophy in postmenopausal women: a randomized, double-blind, placebo-controlled study. Maturitas. 2014 Nov;79(3):316-21. doi: 10.1016/j.maturitas.2014.07.010. Epub 2014 Jul 21. PMID 25104582
- [Background] Labrie F, Archer D, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Berube R, Belanger P, Berger L, Gilbert L, Martel C, Balser J. Serum steroid levels during 12-week intravaginal dehydroepiandrosterone administration. Menopause. 2009 Sep-Oct;16(5):897-906. doi: 10.1097/gme.0b013e31819e8930. PMID 19436226
- [Background] Nachtigall LE. Comparative study: Replens versus local estrogen in menopausal women. Fertil Steril. 1994 Jan;61(1):178-80. doi: 10.1016/s0015-0282(16)56474-7. PMID 8293835
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Erekson EA, Yip SO, Wedderburn TS, Martin DK, Li FY, Choi JN, Kenton KS, Fried TR. The Vulvovaginal Symptoms Questionnaire: a questionnaire for measuring vulvovaginal symptoms in postmenopausal women. Menopause. 2013 Sep;20(9):973-9. doi: 10.1097/GME.0b013e318282600b. PMID 23481118
- See also: Guidance For Industry: Estrogen And Estrogen/Progestin Drug Products To Treat Vasomotor Symptoms And Vulvar And Vaginal Atrophy Symptoms--Recommendations For Clinical Evaluation — https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/ucm071643.pdf